CLINICAL TRIAL: NCT04931485
Title: Protocolised Early De-Resuscitation in Septic Shock (REDUCE) - a Randomised Controlled Multi-centre Feasibility Study
Brief Title: Protocolised Early De-Resuscitation in Septic Shock (REDUCE)
Acronym: REDUCE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REDUCE
Record Dates: First submitted 2021-05-14; First posted 2021-06-18 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Septic Shock
Keywords: Septic shock; Fluid resuscitation
MeSH Terms: conditions — Shock, Septic | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either fluid resuscitation/de-resuscitation according to the REDUCE protocol or standard of care.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: REDUCE Protocol (Experimental): Fluid resuscitation and de-resuscitation is based on the REDUCE fluid management protocol.
  Interventions: Other: Fluid management according to the REDUCE Fluid Protocol
- Standard of Care (Active Comparator): Fluid resuscitation and de-resuscitation according to the standard of care
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Fluid management according to the REDUCE Fluid Protocol — Fluid management according to the protocol will be guided by pre-defined clinical signs for impaired perfusion and fluid overload.
  Other Names: REDUCE protocol
  Arms: Intervention: REDUCE Protocol
Other: Standard of care — Fluid resuscitation and de-resuscitation will be managed according to the standard of care
  Arms: Standard of Care

SUMMARY:
Background: Recent studies have questioned the safety of current fluid resuscitation strategies in patients with septic shock as prospective and observational data suggesting that the resulting fluid overload is associated with mortality. Two strategies have evolved to prevent or minimize fluid overload: restrictive fluid administration or active removal of accumulated fluid. While several small trials show benefits with a restrictive fluid administration regimen, active protocolized de-resuscitation was scarcely evaluated. The combination of both strategies yet warrants systematic evaluation.

Aim: This study aims to assess the efficacy and feasibility of an early active de-resuscitation protocol in patients with septic shock. We hypothesize that the application of a structured early de-resuscitation protocol versus standard of care will lead to less fluid overload at day three after ICU admission.

Study Intervention: Patients admitted to the ICU with confirmed or suspected septic shock (Sepsis-3 definition) will be randomized (1:1) to either the intervention or standard of care. In the intervention arm, patients are managed according to the REDUCE fluid management protocol during resuscitation and de-resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU with the diagnosis of septic shock as defined according to the Sepsis-3 criteria (suspected or confirmed infection AND vasopressor/inotrope ongoing to maintain MAP ≥ 65 mmHg AND Lactate ≥ 2 mmol/l in the last 6 hours

Exclusion Criteria:

* Age <18 years
* Septic shock for more than 12 hours at the time of screening
* Acute burn injury >/= 10% of the body surface area
* Known pregnancy or lactating women
* Consent not obtainable due to national legislation
* Patients on chronic dialysis
* Patients that are known to be allergic to furosemide or metolazone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-05-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patient with a negative fluid balance on day 3 | Up to day 3 after ICU admission
  Proportion of patients with a negative cumulative fluid balance on day 3

SECONDARY OUTCOMES:
Number of patients with fluid overload at day 3 and ICU discharge | From hospital admission to the end of ICU stay, on average after 7 days
  Fluid overload as defined as ((input-output)/admission weight)*100
Feasibility of the REDUCE fluid protocol | From randomisation until the end of ICU stay, on average after 7 days
  Number of REDUCE fluid protocol violations
Incidence of ischemic events and severe AKI | Ischemic events and AKI: From randomisation until the end of ICU stay (on average after 7 days), and at day 30; electrolyte and acid-base/medication associated safety endpoints: during ICU stay (on average 7 days)
  Number of patients with:ischaemic events, severe AKI (AKIN stage 2 or more); respectively episodes of: severe hypernatremia (sodium >/= 155mmol/l), severe hypokalemia (< 3.0 mmol/l), severe metabolic alkalosis (pH >/= 7.55, bicarbonate >/= 35 mmol/l), anaphylactic reaction to diuretic drug
Ventilator-free days at day 30 | Up to 30 days after randomisation
  Ventilator free days up to day 30
Vasopressor-free days at day 30 | Up to 30 days after randomisation
  Vasopressor free days up to day 30
Renal replacement therapy | Up to 90 days after randomisation
  Need for and time on renal replacement therapy
Number of patients with need for renal replacement at 90days | Up to 90 days after randomisation
  Number of patients with on-going need for renal replacement at 90days
All-cause mortality | Up to 90 days after randomisation
  At 30days and 90 days after randomization

OTHER OUTCOMES:
Daily cumulative fluid balance up to day 7 | Throughout the ICU stay, on average 7 days
  Cumulative fluid balance is total input - total output

CONTACTS AND LOCATIONS:
Overall Officials: Anna S Messmer, MD, Principal Investigator — Department of Intensive Care, Inselspital, Bern University Hospital, Bern, Switzerland
Locations (4):
- Switzerland (4):
  - University Hospital Basel, Basel
  - University Hospital Bern, Inselspital, Bern
  - Cantonal Hospital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Messmer A, Pietsch U, Siegemund M, Buehler P, Waskowski J, Muller M, Uehlinger DE, Hollinger A, Filipovic M, Berger D, Schefold JC, Pfortmueller CA. Protocolised early de-resuscitation in septic shock (REDUCE): protocol for a randomised controlled multicentre feasibility trial. BMJ Open. 2023 Sep 21;13(9):e074847. doi: 10.1136/bmjopen-2023-074847. PMID 37734896